CLINICAL TRIAL: NCT05649527
Title: Nutri-Bébé 2022 A French National Survey on Feeding Practice and Nutrient Intakes of Children Under 3 Years of Age
Acronym: NBB2022
Status: Completed | Type: Observational
Sponsor: Secteur Français des Aliments de l'Enfance (Industry)
Collaborators: IPSOS (Industry); Centre de Recherche pour l'Etude et l'Observation des Conditions de Vie (Unknown)
Responsible Party: Sponsor
Other Study IDs: NBB 2022; QD0300 (Other Grant/Funding Number: Secteur Français des Aliments de l'Enfance (SFAE)); 2020-A03538-31 (Registry Identifier: Research registration ID (ID RCB))
Record Dates: First submitted 2022-12-02; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Feeding Behavior; Nutrients Intakes
Keywords: Nutrition survey; Feeding practice; Nutrients intake; Infant; Toddler
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main sample: Sample of 880 children spontaneously recruited and representative of the French population according to the criteria defined for the study. Includes breastfed children.
- Additional sample: Children in the appropriate age group selected because of their specific consumption in order to increase the number of children in the concerned age group to allow a statist test.

SUMMARY:
The Nutri-Bébé 2022 survey is an observational cross-sectional study aiming to update food consumption, practices and nutrient intakes in children under 3 years of age in metropolitan France.

DETAILED DESCRIPTION:
Infant's and young children's diet is a determining factor in their growth and development and may impact the occurrence of non-communicable diseases in the medium and long term. In this context, knowledge regarding the feeding practice and nutrients intake in children under 3 years of age is valuable, whether for the entire scientific and medical community or for the public authorities.

Aiming to help achieving this objective, the SFAE has carried out a national observational survey every 8 years since 1981. The analysis of these data over time makes it possible to evaluate the intakes of different nutrients, to note possible nutritional insufficiencies or excesses, potentially linked to bad eating habits. On these bases, this repeatable survey can alert health professionals and help refine public health nutrition policy in France. A new edition was launched between March 2022 and July 2022 by an official polling institute, IPSOS. The sample includes more than 1,200 children aged from 0.5 to 35 months, distributed in 11 age-groups of equal importance, and living in metropolitan France (excluding Corsica).

This is a cross-sectional observational survey.

IPSOS fulfills the following standards and industry requirements (ESOMAR professional code of conduct and standards, ISO 20252:2012 international standard for market, opinion and social research, French data protection act (loi "informatique et libertés "). IPSOS ensures to conduct the surveys in accordance with the regulation on personal data protection and that respondents' personal identity is withheld. The SFAE has undertaken with the "Commission Nationale de l'Informatique et des Libertés" (CNIL), the French data protection authority) to respect the MR-003 reference methodology and is authorized to set up the processing of data without prior authorization from the CNIL (declaration n° 2220501 of 2020/12/18).

Information on the children will be collected directly from the responding parents (primarily responsible for their child's diet). The collection of information will be carried out according to the following successive stages:

* recruitment of families according to the quota method, provided they are fluent in French language and can use a computer.
* To be included children should be born at term with a birth weight ≥ 2500 g and should have no intercurrent acute or chronic disease.
* Face-to-face interview at home by an investigator to collect informed consent of the parents, sociodemographic data, child weight and height as well as information on children's eating habits.
* Completion by the parent of an online consumption diary for a period of 3 non-consecutive days (2 weekdays and 1 weekend day, with at least one day of separation between each collection day).
* Self-questionnaire to be completed by the responding parent on the child's diet, context and physical activities.

The study conducted in 2022 is the sixth edition of the Nutri-Bébé survey.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 0.5 to 35 months
* Child whose responding parent, mainly responsible for his diet, agrees to complete the three stages of the survey (informed consent).
* Child whose responding parent accepts the collection of birth weight, and the most recent weight and height in the health booklet. If the weight measurement has not been performed recently, the responding parent agrees to measure the weight of their child during the first interview. In this case, the presence of the child will be necessary. A recent weight corresponds to a measurement in the 15 days preceding inclusion for children aged 0-6 months, in the month preceding inclusion for children aged 6-12 months and in the two months preceding inclusion for those over one year old.
* Child whose parents have been informed of the study orally and in writing, and have not objected to the participation of the child before its inclusion and to the collection of information concerning them.
* In the case of the spouse of the responding parent, different from the second parent and living in the same household, no opposition to the collection of data concerning him

Exclusion Criteria:

* Child with a chronic or intercurrent pathology (including food allergies)
* Child with a birth weight of less than 2.5 kg
* Child whose last weight measurement in the health record is not recent enough AND whose parent refuses to measure his weight
* Child having to take at least one meal at school during the 3 days of filling in the consumption diary
* Child cared for by the crèche or by a third party and whose person responsible for meals refuses to send all the information (qualitative and quantitative) to the responding parent so that he can complete the consumption diary
* Child whose sponsoring parent is under the age of 18, or is placed under guardianship or curatorship, or under legal protection

Ages: 15 Days to 35 Months | Sex: All
Age Groups: Child
Study Population: Children from 0.5 to 35 months old, residing in metropolitan France.
Sampling Method: Probability Sample
Enrollment: 1224 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Age at inclusion | March to July 2022
  months
Weight | March to July 2022
  kg
Height | March to July 2022
  cm
Prevalence of children breastfed | March to July 2022
  frequency in %
Prevalence of children formula-fed | March to July 2022
  frequency in %
introduced complementary food specific baby food and adult type food | March to July 2022
  frequency in %
Age at introduced complementary food | March to July 2022
  months
Mean over 3 days of Food quantities | March to July 2022
  g/day
Mean over 3 days of macronutrient intake (protein, lipid, carbohydrate, fiber) | March to July 2022
  g/d
Mean over 3 days of Intakes of Linoleic-, alpha linolenic-acids, DHA, ARA, minerals (sodium, calcium, phosphorus, magnesium, iron, zinc), Vitamin B1,B2, B3, B6, C, E | March to July 2022
  mg/d
Mean over 3 days of intakes of Vitamin B9, B12, Retinol, Beta-caroten | March to July 2022
  µg/d
Vitamin A intake | March to July 2022
  RE(Retinol Equivalent)/d

SECONDARY OUTCOMES:
Influence of parents professional activity data on practice | March to July 2022
  p value Scale : professions and socio-professional categories (PCS) minimum: inactive maximum: high socio-professional categories (executives and higher intellectual professions)
Influence of economic status on practice | March to July 2022
  p value Household income scale Minimum : <1700€/months Maximum : >5400€/months
Influence of level of education on practice | March to July 2022
  p value 3 level scale minimum: Primary or secondary education maximum: Higher education
Duration of previous breastfeeding | March to July 2022
  months

OTHER OUTCOMES:
Previous feeding | March to July 2022
  Frequency in % of type of formula previously used
Screen exposure | March to July 2022
  frequency in % of exposure to screens at different times of consumption
Screen exposure | March to July 2022
  minutes/day spent in front of a screen
Physical activity | March to July 2022
  minutes/day

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre CHOURAQUI, MD, MSc, Principal Investigator — Pediatric depart. Gastroenterology and Nutrition division University Hospital Grenoble-Alpes France; Amandine ROCHEDY, PhD, Principal Investigator — UTM Department of Sociology and Anthropology. University Toulouse - Jean Jaurès ;; Sandra BRANCATO, MD, Principal Investigator — Medical practice, Brignon; Domitille HERMITE, MSc, Principal Investigator — IPSOS; Mathilde GRESSIER, MSc, Principal Investigator — CREDOC; Virginie SOMON, Engineer,MSc, Study Director — Secteur Français des Aliments de l'Enfance
Locations (1):
- IPSOS, Paris, France

IPD SHARING:
Plan to Share IPD: No
To be shared is the global report of results on each items (food practices, food consumption, nutrients intakes), according to age groups.

REFERENCES:
- [Background] Chouraqui JP, Tavoularis G, Emery Y, Francou A, Hebel P, Bocquet M, Hankard R, Turck D. The French national survey on food consumption of children under 3 years of age - Nutri-Bebe 2013: design, methodology, population sampling and feeding practices. Public Health Nutr. 2018 Feb;21(3):502-514. doi: 10.1017/S1368980017002518. Epub 2017 Nov 2. PMID 29094670
- [Background] Chouraqui JP, Tavoularis G, Simeoni U, Ferry C, Turck D. Food, water, energy, and macronutrient intake of non-breastfed infants and young children (0-3 years). Eur J Nutr. 2020 Feb;59(1):67-80. doi: 10.1007/s00394-018-1883-y. Epub 2019 Jan 16. PMID 30648220
- [Background] Chouraqui JP, Tavoularis G, Turck D, Ferry C, Feillet F. Mineral and vitamin intake of infants and young children: the Nutri-Bebe 2013 survey. Eur J Nutr. 2020 Sep;59(6):2463-2480. doi: 10.1007/s00394-019-02093-3. Epub 2019 Sep 25. PMID 31555975
- [Background] Chouraqui JP, Turck D, Tavoularis G, Ferry C, Dupont C. The Role of Young Child Formula in Ensuring a Balanced Diet in Young Children (1-3 Years Old). Nutrients. 2019 Sep 13;11(9):2213. doi: 10.3390/nu11092213. PMID 31540250
- [Background] Chouraqui JP, Darmaun D, Salmon-Legagneur A, Shamir R. Protein intake pattern in non-breastfed infants and toddlers: A survey in a nationally representative sample of French children. Clin Nutr. 2022 Feb;41(2):269-278. doi: 10.1016/j.clnu.2021.12.006. Epub 2021 Dec 8. PMID 34998033
- [Background] Chouraqui JP, Thornton SN, Seconda L, Kavouras SA. Total water intake and its contributors in infants and young children. Br J Nutr. 2022 Aug 14;128(3):531-541. doi: 10.1017/S0007114521003469. Epub 2021 Sep 9. PMID 34496987